CLINICAL TRIAL: NCT02421575
Title: Assessment of the Biological Effect of Autophagic Inhibition With Hydroxychloroquine in Prostate Cancer
Brief Title: Hydroxychloroquine in Blocking Autophagy in Patients With Prostate Cancer Undergoing Surgery or Active Surveillance
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 121102; NCI-2014-02216 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0220110278; 121102 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2014-12-10; First posted 2015-04-20 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group I, Arm I (lower dose hydroxychloroquine) (Experimental): Patients receive hydroxychloroquine PO QD for 14 days and then undergo prostatectomy.
  Interventions: Drug: Hydroxychloroquine; Other: Laboratory Biomarker Analysis
- Group I, Arm II (higher dose hydroxychloroquine) (Experimental): Patients receive hydroxychloroquine PO TID for 14 days and then undergo prostatectomy.
  Interventions: Drug: Hydroxychloroquine; Other: Laboratory Biomarker Analysis
- Group II (mid-dose hydroxychloroquine) (Experimental): Patients receive hydroxychloroquine PO QD. Treatment continues until the beginning of local therapy or for up to 1 year.
  Interventions: Drug: Hydroxychloroquine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Hydroxychloroquine — Given PO
  Other Names: HCQ
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase 0 trial studies hydroxychloroquine in blocking autophagy in patients with prostate cancer who are undergoing surgery or active surveillance. Autophagy is a process in which cells break down some parts of themselves to stay alive during times of stress, such as starvation. This may allow cancer cells to survive damage from chemotherapy. Hydroxychloroquine may block this process from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of different doses of hydroxychloroquine on markers of autophagy in prostate tumor.

SECONDARY OBJECTIVES:

I. To determine the distribution of autophagic activity within prostate cancer tissue.

II. To determine the utility of beclin-1 as a marker of autophagic activity. III. To assess markers of apoptosis in tumor tissue. IV. To perform deep-sequencing on prostate tissue obtained at the time of surgery.

V. To assess prostate-specific antigen (PSA) as a biochemical endpoint of clinical activity.

VI. To determine the number of circulating tumor cells (CTCs) in pre- and post-treatment blood samples.

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP I (PLANNING PROSTATECTOMY): Patients in Group I are randomized to 1 of 2 arms.

ARM I: Patients receive hydroxychloroquine orally (PO) once daily (QD) for 14 days and then undergo prostatectomy.

ARM II: Patients receive a higher dose of hydroxychloroquine PO thrice daily (TID) for 14 days and then undergo prostatectomy.

GROUP II (ACTIVE SURVEILLANCE): Patients receive hydroxychloroquine PO QD. Treatment continues until the beginning of local therapy or for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Have abnormal digital rectal examination, or abnormal prostate specific antigen (> 4.0 ng/ml), or obstructing prostate, or biopsy proven prostate cancer
* Scheduled for prostate surgery, i.e. transurethral resection of the prostate (TURP) or prostatectomy
* Planned to be treated by active surveillance

Exclusion Criteria:

* Patients on treatment for rheumatoid arthritis or systemic lupus erythematosus
* Patients with psoriasis
* Patients receiving any disease-modifying anti-rheumatic drug (DMARD)
* Active clinically significant infection requiring antibiotics
* Patients with glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Patients taking other commercially available medications which may theoretically either stimulate or inhibit autophagy, which are calcitriol and chloroquine
* Patients taking medications which may lead to interactions with hydroxychloroquine, including penicillamine, telbivudine, botulinum toxin, digoxin, and propafenone
* Patients must not have prior visual field changes from prior 4-aminoquinoline compound use
* Must not be taking hydroxychloroquine for treatment or prophylaxis of malaria
* History of hypersensitivity to 4-aminoquinoline compound

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-07; Primary Completion 2016-02-26 (Actual); Study Completion 2016-02-26 (Actual)

PRIMARY OUTCOMES:
Change in markers of autophagy in prostate tumor (Group I) | Baseline to 14 days (time of surgery)
Levels of markers of autophagy in prostate tumor (Group II) | Up to 1 year

SECONDARY OUTCOMES:
Distribution of autophagic activity in prostate cancer tissue | Up to 1 year
Autophagic activity, assessed by beclin-1 levels | Up to 1 year
  The utility of beclin-1 as a marker of autophagic activity will be determined.
Levels of markers of apoptosis in tumor tissue | Up to 1 year
Clinical activity, as assessed by PSA levels | Up to 1 year
Number of CTCs in blood samples | Up to 1 year
  The number of CTCs in pre- and post-treatment blood samples will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Singer, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States